CLINICAL TRIAL: NCT05787223
Title: Effects of Balance Training Exercises on Mobility in Open and Closed Environment in Children With Visual Impairments.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0705
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator)
  Interventions: Other: Baseline Treatment
- Experimental Group (Experimental)
  Interventions: Other: Baseline Treatment; Other: Dynamic Training

INTERVENTIONS:
Other: Baseline Treatment — Control Group that will be provided with be given baseline treatment of static balance training (static exercise like standing on balance board, bounce on one foot, heel rises/toe rises, standing on one foot, jumping on trampoline)
Other: Dynamic Training — Experimental Group that will be provided with base line treatment along with dynamic balance training (cross, side &tandem walking, step up and down, jumping &hopping on floor). Exercises Will be given the 40 minutes with 2 sessions per week over the period of 08 weeks
  Arms: Experimental Group

SUMMARY:
Visual impairment is used to describe any kind of vision loss, whether it's someone who cannot see at all or someone who has partial vision loss. Visual impairment is classified on the basis of visual acuity like mild, moderate, severe, profound, near total visual impairment, no light perception (NLP). Balance is defined as the ability to maintain one's equilibrium as the center of gravity when the COG shifts called (dynamic balance), as in walking and running, and while the center of gravity remains stationary (static balance). Mobility is the ability of a patient to change and control their body position. Physical mobility requires sufficient muscle strength and energy, along with adequate skeletal stability, joint function, and neuromuscular synchronization. This will be a randomized controlled trial. Approval will be gained from the Ethical committee of the Riphah international university Lahore, Pakistan prior to the commencement of study. Written informed consent will be taken from all the patients and all information and data will be confidential. Subjects will be informed that there is no risk of study and they will be free to withdraw any time during process of study. 24 patients will be divided into two Groups. Group A will be the Control Group that will be given the baseline treatment of static balance training (static exercises like standing on balance board, bounce on one foot, heel rises/toe rises, standing on one foot, jumping on trampoline) and Group B will be the Experimental Group that will be provided with baseline treatment along with dynamic balance training (cross, side and tandem walking, step up and down, jumping and hopping on floor). Exercises will be given the 40 minutes with 2 sessions per week over the period of 8 weeks. Pre and Post treatment values will be evaluated. The tools used will be Time Up and Go Test, GMFM-88, Wee FIM. Data will be analyzed using SPSS 22.0 and mean and standard deviation will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* 08-14 Age
* Visual acuity is 20/70 with possible correction
* All participants are label with legally blind by an ophthalmologist.
* Able to follow the commands

Exclusion Criteria:

* Those who were unable to complete follow-up tests.
* No other neurological or orthopedic problems that could affect balance, and who could understand the instructions during the implementation of the exercises and tests.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Time Up and Go Test | Baseline and 8th week
  The Timed Up and Go (TUG) test is a performance-based measure of functional mobility that was initially developed to identify mobility and balance impairments in older adults
Gross Motor Function Measure (GMFM-88) | Baseline and 8th week
  The Gross Motor Function Measure31 is a criterion-referenced assessment designed to be used with children with cerebral palsy. It evaluates the child's ability to complete motor functions, such as rolling, crawling, sitting, standing, walking, running, stair use, and jumping. A four-point ordinal scale of measurement is used to assess each item. A score of 0 indicates the task cannot be done, 1 indicates the task can be initiated (<10% completion), 2 indicates partial completion of the task (10% to <100% completion), and 3 indicates the task can be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute for Special Children, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ackland P, Resnikoff S, Bourne R. World blindness and visual impairment: despite many successes, the problem is growing. Community Eye Health. 2017;30(100):71-73. No abstract available. PMID 29483748
- [Background] Parreira RB, Grecco LAC, Oliveira CS. Postural control in blind individuals: A systematic review. Gait Posture. 2017 Sep;57:161-167. doi: 10.1016/j.gaitpost.2017.06.008. Epub 2017 Jun 12. PMID 28641161
- [Background] Winnick JP. The Performance of Visually Impaired Youngsters in Physical Education Activities: Implications for Mainstreaming. 1985;2(4).
- [Background] Behar MP, Zucker DRJJoVI, Blindness. Sensory Awareness Exercises for the Visually Handicapped. 1976;70(4):146-8.
- [Background] Lewis V, Norgate S, Collis G, Reynolds RJBJoDP. The consequences of visual impairment for children's symbolic and functional play. 2000;18(3):449-64.